CLINICAL TRIAL: NCT02343276
Title: Randomized Clinical Trial Comparing Transradial Catheterization With or Without Spasmolytic Drugs.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Cardiologia de Santa Catarina (Other)
Responsible Party: Principal Investigator, Roberto Léo da Silva, MD, Instituto de Cardiologia de Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ICSC-2015
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-02

CONDITIONS: Cardiac Catheterisation
Keywords: Radial Spasm
MeSH Terms: conditions — Spasm | interventions — Nitroglycerin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (saline solution 10 ml) in radial artery after sheath insertion
  Interventions: Other: Placebo
- Intervention (Experimental): Nitroglycerin (200 micrograms) + saline solution 10 ml in radial artery after sheath insertion
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — Nitroglycerin (200 micrograms) + saline solution 10 ml in radial artery after sheath insertion
  Other Names: Tridil
  Arms: Intervention
Other: Placebo — Placebo (saline solution 10 ml) in radial artery after sheath insertion
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
Single-center study, randomized, double-blind, placebo controlled, with patients undergoing diagnostic or therapeutic catheterization via the transradial approach. Patients will be randomized into two groups: one group will receive the vasodilator nitroglycerin during the procedure (intervention group), and a second group will receive saline 0.9% in the same volume and time during the procedure (control group).

Will be evaluated: incidence of spasms of the radial artery, ability to perform the procedure without the need to change the access site, pain presented by the patient, time and total radiation of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac catheterization
* Suitable candidates for transradial approach

Exclusion Criteria:

* AMI
* Intubated patients
* Complications during procedure (cardiac arrest, pulmonary edema, cardiogenic shock, stroke)
* Prior inclusion in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto L da Silva, MD, Principal Investigator — Instituto de Cardiologia de Santa Catarina
Locations (1):
- Instituto de Cardiologia de Santa Catarina, São Jose, Santa Catarina, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was designed as a single-centre, prospective, randomised, placebo-controlled, double-blind trial with an all-comers design. All eligible patients were aged 18 years or over with a clinical indication for coronary angiography (ad hoc angioplasty was allowed) or percutaneous coronary intervention (PCI).
Period: Overall Study
Arm/Group | Placebo | Intervention
Started | 164 | 164
Completed | 164 | 164
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Intervention | Total
Number analyzed (Participants) | 164 | 164 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.79 (11.15) | 60.93 (11.90) | 60.36 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 116
  Male | 106 | 106 | 212
Region of Enrollment [Number; unit: participants]
  Brazil | 164 | 164 | 328
Height [Mean (Standard Deviation); unit: METERS] | 1.65 (0.09) | 1.64 (0.09) | 1.65 (0.09)
Weight [Mean (Standard Deviation); unit: KILOGRAMS] | 76.61 (28.13) | 76.59 (28.47) | 76.6 (28.24)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.13 (7.33) | 28.47 (7.45) | 28.32 (7.41)

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment Using Visual Analogue Scale
Description: the patients' feeling of pain in the forearm, and it was measured using a visual analogue scale (VAS), applied at the end of the procedure by an interventional nurse. The VAS consists of a single line measuring 100 mm, anchored by verbal descriptors, saying 'no pain' and 'worst possible pain'. Higher values mean a worse pain.
Time Frame: Five minutes after sheath removal
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 164 | 164
score on a scale | 24.75 (23.1) | 24.74 (26.0)

2. Secondary Outcome: Procedure Duration
Description: Procedure duration, from artery catheterization up to removal of sheath.
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 164 | 164
minutes | 22.24 (12.31) | 21.36 (13.57)

3. Secondary Outcome: Radiation Exposure
Description: Total radiation required to complete the procedure.
Time Frame: Immediate
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Placebo | Intervention
Number analyzed (Participants) | 164 | 164
mGy | 660.92 (433.25) | 655.61 (441.64)

ADVERSE EVENTS:
Arm/Group | Placebo | Intervention
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/164
Other Adverse Events (participants affected / at risk) | 0/164 | 0/164

LIMITATIONS AND CAVEATS:
Procedures were conducted in a single, high-volume center. All, but one, operators had high experience in radial access.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No